CLINICAL TRIAL: NCT05279937
Title: The Use of Ultrasound-Guided Dextrose Prolotherapy in Low Back Pain in Patients With Hypermobile-Type, Ehlers-Danlos Syndrome
Brief Title: The Ultrasound-Guided Dextrose Prolotherapy in Ehlers-Danlos Syndrome Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-380
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Ehlers-Danlos Syndrome; Low Back Pain; Sacroiliac Instability
Keywords: Prolotherapy; Dextrose; Ultrasound
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Low Back Pain | interventions — Glucose; Lidocaine

STUDY DESIGN:
Intervention Model Description: 10mL of 1% Lidocaine (Control) or 5mL of 50% Dextrose + 5mL of 1% Lidocaine (Prolotherapy).
Who Masked: Participant, Investigator
Masking Description: Double blinded randomized
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prolotherapy (Experimental): 5mL of 50% Dextrose + 5mL of 1% Lidocaine (Prolotherapy).
  Interventions: Drug: Dextrose 50% Intravenous Solution
- Control (Active Comparator): 10mL of 1% Lidocaine (Control)
  Interventions: Drug: Lidocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Dextrose 50% Intravenous Solution — 5mL of 50% Dextrose + 5mL of 1% Lidocaine (Prolotherapy).
  Arms: Prolotherapy
Drug: Lidocaine 1% Injectable Solution — 10mL of 1% Lidocaine (Control)
  Arms: Control

SUMMARY:
1. Specific Aim: To show the safety and efficacy of prolotherapy injection for chronic sacroiliac and myofascial lumbar pain while standardizing an ultrasound guided injection technique
2. Specific Aim: To demonstrate that dextrose prolotherapy subjectively decreases lumbar back pain (LBP) associated with chronic sacroiliac (SI) and myofascial lumbar back pain/injury in patients with Hypermobile-Type Ehlers-Danlos Syndrome (hEDS).
3. Specific Aim: To use ultrasound (US) guidance to identify SI and myofascial lumbar back pain/injury for targeted dextrose prolotherapy treatment and to provide objective measures of decreasing inflammation via Power Doppler and ligament repair.
4. Specific Aim: To determine if US-guided dextrose prolotherapy decreases the direct costs of care for chronic LBP in contrast to conventional therapies by reducing return visits, specialty referrals, physical therapy, medications, and unnecessary procedures.

DETAILED DESCRIPTION:
The goal of this research project is to prove that ultrasound-guided prolotherapy is a cost effective and curative treatment option for chronic low back pain in Hypermobile-Type Ehlers-Danlos Syndrome (hEDS). Ultrasound (US) will be used to assist in proper evaluation of the thoracolumbar fascial complex (TLFC), long posterior sacroiliac ligament (LPSL), multifidi and gluteus maximus along with precise administration of medication into identified regions of interest. By comparing targeted lidocaine and concentrated dextrose (prolotherapy) injections, placebo effect or therapeutic local trauma created by the needle, like dry needling can be ruled out. The combination of subjective data collection with Owestry Disability Index (ODI) and the Number Rating Scale (NRS) assessments and objective findings on ultrasound imaging such as Pixel Ratio and ligament integrity will provide sufficient information to determine if prolotherapy is effective at reducing inflammation, providing prolonged pain relief, and return to function in patients with hEDS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-75
* Subjects who resent to Tulane Institute of Sports Medicine and Tulane Lakeside with low back pain that is diagnosed as chronic (>3 months) SI dysfunction or myofascial lumbar pain with a diagnosis of hEDS per The International Consortium on Ehlers-Danlos Syndrome and Related Disorders diagnostic criteria.
* Diagnosis will include but not be limited to physical exam findings consistent with tenderness to palpation over the sacroiliac joint (SIJ) or posterior superior iliac crest, and upper outer quadrant of the gluteus maximus.
* Diagnosis will also include US-guided tenderness to palpation of the thoracolumbar facial complex insertion into the posterior superior iliac spine (PSIS), SI, or gluteus maximus.
* Further testing will include US evaluation using a General Electric Logiq E ultrasound machine to look for any evidence of structural abnormality or reactive hyperemia of the TLFC, LPSL, multifidus or gluteus maximus.

Exclusion Criteria:

* Patients >75 and < 18 years old.
* Any patient with evidence of lumbar radiculopathy, acute lower back pain, pregnancy, prior lumbosacral surgery, opiate use within the last 6 months, steroid exposure within 6 weeks, NSAID exposure within 2 weeks.
* Patients who are unwilling to stop taking or admit to receiving NSAIDs or any form of corticosteroids during the study.
* Patients with a history of bleeding disorders, severe thrombocytopenia, immunodeficiency disorder, and hypersensitivity of local anesthetics of amide type will be excluded along with any patient who actively has systemic bacterial infection with fever, skin infection over the injection site, or takes anti-platelet/anti-coagulant medication.
* Patients with comorbidities such as diabetes mellitus, rheumatoid arthritis, lupus, or any other condition that increases risk of infection may be excluded from the study pending severity and current treatment of their condition.
* Patients receiving workers compensation, disability or who are involved in litigation will also be excluded due to risk of secondary gain.
* Physical exam findings, X-rays, and US imaging will be utilized to determine eligibility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measuring the functionality of the lumbar spine by using Oswestry Low Back Pain Disability Questionnaire in patients with Hypermobile-Type Ehlers-Danlos Syndrome (hEDS) | 12 Months
  The functionality of the lumbar spine will be measured by Oswestry Low Back Pain Disability Questionnaire, which is a tool to measure a patient's permanent functional disability. Each patient uses the questioner the first time they are in clinic and then in each of the follow up visits post treatment until the study completion. The questioner determines if the patient has sustained clinical improvement. The higher the score the more severe low back pain is.

SECONDARY OUTCOMES:
Measuring the change of low back pain via the number rating scale in patients with Hypermobile-Type Ehlers-Danlos Syndrome (hEDS) | 12 Months
  The change in low back pain will be measured by the number rating scale, which is a scale from 1 to 10 measuring low back pain. The higher the score the more severe the pain is in the low back.
The measure of soft tissue inflammation via ultrasound in patients with Hypermobile-Type Ehlers-Danlos Syndrome (hEDS) | 12 Months
  Inflammation will be measured by Doppler ultrasound to determine the degree of inflammation in the area of interest which is measured as Pixel Ration (PR) to show if there is a change or decrease of inflammation with prolotherapy treatment.
The measure of ligament integrity via ultrasound in patients with Hypermobile-Type Ehlers-Danlos Syndrome (hEDS) | 12 Months
  Ligament Integrity will be measured by ultrasound, which will be used to evaluate the quality of ligamentous structures before and after prolotherapy treatment to determine if prolotherapy has the ability to promote tissue regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Courseault, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane Hospital and Clinics, New Orleans, Louisiana, United States